CLINICAL TRIAL: NCT03931473
Title: Efficacy of Two Dual Active Ingredient Long Lasting Insecticidal Nets for Control of Malaria Transmitted by Pyrethroid Resistant Vectors in Benin
Acronym: NNP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: London School of Hygiene and Tropical Medicine (Other)
Collaborators: Centre de Recherche Entomologique de Cotonou (Unknown); UNITAID (Other); Innovative Vector Control Consortium (Unknown); Global Fund (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: NewNetsProject
Record Dates: First submitted 2019-04-25; First posted 2019-04-30 (Actual); Last update posted 2024-10-18 (Actual); Status verified 2024-10

CONDITIONS: Malaria; Anemia
Keywords: Long Lasting Insecticidal Net, Chlorfenapyr, Pyriproxyfen, Pyrethroid, Randomised Controlled Trial, Benin, Vector Control, Malaria
MeSH Terms: conditions — Malaria; Anemia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Interceptor G2 (Experimental): Chlorfenapyr/alpha-cypermethrin
  Interventions: Other: Bed nets
- Royal Guard (Experimental): Pyriproxyfen/alpha-cypermethrin
  Interventions: Other: Bed nets
- Interceptor (Active Comparator): Alpha-cypermethrin
  Interventions: Other: Bed nets

INTERVENTIONS:
Other: Bed nets — Next-generation bed nets combining insecticides with different modes of action or a standard pyrethroid bed net

SUMMARY:
The massive scale-up of Long Lasting Insecticidal Nets (LLIN) has led to a major reduction in malaria burden (up to 50%) in many sub-Saharan African countries. This progress is threatened by the wide scale selection of insecticide resistant malaria vectors. New types of LLIN combining a mixture of two insecticides have been developed to control resistant mosquitoes.

The efficacy of two bi-treated LLIN are compared to a standard LLIN in a three-arm, single blinded, cluster-randomized trial in Cove, Benin. The arms are; 1/ Royal Guard, a net combining pyriproxyfen (PPF), which is known to disrupt female reproduction and fertility of eggs, and the pyrethroid alpha-cypermethrin, 2/Interceptor G2, LLIN incorporating a mixture of two adulticides with different modes of action; chlorfenapyr and a pyrethroid (alpha-cypermethrin), and 3/ The control arm: Interceptor, a standard LLIN treated with alpha-cypermethrin.

The primary outcome of the trial will be malaria case incidence in children aged 6 months to 10 years.

DETAILED DESCRIPTION:
Background: The massive scale-up of Long-Lasting Insecticidal Nets (LLIN) has led to a major reduction in malaria burden (up to 50%) in many sub-Saharan African (SSA) countries. This progress is threatened by the wide scale selection of insecticide resistant malaria vectors.

Study site: The study will be conducted in the districts of Cove, Zagnanado and Ouinhi, a collection of three districts found in the Zou department in Benin. This area consists of 100 villages with approximately 40,000 households and a population size of 191,000.

The aim of this research is to evaluate the efficacy of 2 novel dual active Ingredient (AI) LLINs in a community randomized controlled trial on epidemiology outcomes. The trial will take place over 2 years in an area where malaria vectors are resistant to pyrethroid insecticide in Benin, West Africa. Update- the trial is now continuing for a third year.

The primary objective is to assess the efficacy of next generation LLIN on malaria case incidence in children aged 6 months to 10 years, compared to standard LLINs. The secondary objectives are to evaluate the efficacy of the 2 bi-treated LLIN as compared to standard LLIN on a) malaria infection prevalence in children aged 6 months to 10 years; b) prevalence of moderate and severe anaemia in children under 5 years old and c) entomological inoculation rate (EIR) (as a proxy for malaria transmission). In addition, we will compare potential insecticide resistance selection, between the 3 trial arms and evaluate the impact of the new types of LLIN on other entomological outcomes (species composition, blood feeding, resting/feeding behaviour and sterility (oocyte [egg] development).

Study design: Three-arm superiority, single blinded, cluster-randomized trial with village as the unit of randomisation. The arms consist of; 1/ Royal Guard, a net combining pyriproxyfen (PPF), which is known to disrupt female reproduction and egg fertility, and the pyrethroid alpha-cypermethrin, 2/Interceptor G2, a mixture LLIN incorporating two adulticides with different modes of action; chlorfenapyr and a pyrethroid (alpha-cypermethrin), and 3/ The control arm: Standard LLIN Interceptor is an alpha-cypermethrin only LLIN.

The primary outcome of the trial will be incidence of malaria cases (confirmed by rapid diagnostic test (RDT)) in children aged 6 months to 10 years followed for 24 months. Update: the study is now continuing for a further year.

Secondary outcomes are cross-sectional community prevalence of malaria infection (confirmed by RDT) in the study population at 6- and 18-months post-intervention, prevalence of moderate and severe anaemia in children under 5 years old, entomological inoculation rates (EIR), vector density and insecticide resistance intensity. Update: there will also be a 30 month cross-sectional survey.

Sample size: To compare incidence of malaria cases between study arms, we will recruit a cohort of 25 children per cluster in 60 clusters for 24 months follow up to be able to detect a 30% relative reduction in malaria cases per child per year (rate ratio 0.7) between the intervention and the reference arms. The children will be visited twice a month during the transmission season (April to November) and once a month during the dry season. We will conduct malaria infection prevalence cross-sectional surveys, at 6 and 18 months after LLIN distribution. 40 households will be randomly selected from each of the 60 clusters (20 clusters per arm x 3 arms) and information on education, socio economic status, LLIN ownership and usage recorded during each survey. From these 40 households per cluster we will randomly select 70 individuals. The study will have 80% power to detect a relative 30% lower prevalence (prevalence ratio 0.70 in each intervention arm (Royal Guard or Interceptor G2) relative to standard LLIN. Entomological inoculation rate (EIR) will be measured bi-monthly for 2 years in 8 households per cluster in all the clusters. Update: Follow up for cohort children was suspended during the pandemic meaning the primary outcome only included 21 months of follow up- to counteract this, 30 children were selected in each cluster. The follow up is now continuing up to 36 months- post-distribution. Due to logistics, the entomological data collection took place in 4 houses in each cluster every 3 months.

Frequency and intensity resistance assay with An. gambiae, An. arabiensis and An.funestus will be performed using permethrin, alpha-cypermethrin, pyriproxyfen and chlorfenapyr in 6 clusters (2 clusters per arm). An. gambiae s.l. and An. funestus will be screened for mutations in insecticide target sites (Vgsc) and metabolic resistance following CYp6 genes a small group of P450s that are over expressed in insecticide resistant populations. Changes in frequency of these genes and target site mutation will be followed every year in the three arms.

ELIGIBILITY:
Inclusion Criteria for cohort:

* Children aged 6 months to 9 years
* Resident in study villages
* Written, informed consent from guardians

Exclusion Criteria:

* Non-residents

Ages: 6 Months to 9 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1800 (Actual)
Dates: Start 2020-06-01 (Actual); Primary Completion 2023-05-01 (Actual); Study Completion 2023-05-01 (Actual)

PRIMARY OUTCOMES:
Malaria Case Incidence | 2 years
  Malaria case incidence in children aged 6 months to 10 years measured through bi-monthly/monthly visits

SECONDARY OUTCOMES:
Malaria Infection prevalence | 18 months
  Malaria infection prevalence measured in cross-sectional surveys 6 months and 18 months post- distribution
Entomological Inoculation Rate | 2 years
  EIR measured every quarter during entomological surveys

CONTACTS AND LOCATIONS:
Overall Officials: Martin C Akogbéto, PhD, Principal Investigator — Centre de Recherche Entomologique de Cotonou; Natacha Protopopoff, PhD, Principal Investigator — London School of Hygiene and Tropical Medicine
Locations (1):
- Manfred Accrombessi, Cové, Benin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Accrombessi M, Cook J, Ngufor C, Sovi A, Dangbenon E, Yovogan B, Akpovi H, Hounto A, Thickstun C, Padonou GG, Tokponnon F, Messenger LA, Kleinschmidt I, Rowland M, Akogbeto MC, Protopopoff N. Assessing the efficacy of two dual-active ingredients long-lasting insecticidal nets for the control of malaria transmitted by pyrethroid-resistant vectors in Benin: study protocol for a three-arm, single-blinded, parallel, cluster-randomized controlled trial. BMC Infect Dis. 2021 Feb 19;21(1):194. doi: 10.1186/s12879-021-05879-1. PMID 33607958
- [Background] Yovogan B, Sovi A, Padonou GG, Adoha CJ, Akinro B, Chitou S, Accrombessi M, Dangbenon E, Akpovi H, Messenger LA, Osse R, Hounto AO, Cook J, Kleinschmidt I, Ngufor C, Rowland M, Protopopoff N, Akogbeto MC. Pre-intervention characteristics of the mosquito species in Benin in preparation for a randomized controlled trial assessing the efficacy of dual active-ingredient long-lasting insecticidal nets for controlling insecticide-resistant malaria vectors. PLoS One. 2021 May 20;16(5):e0251742. doi: 10.1371/journal.pone.0251742. eCollection 2021. PMID 34014982
- [Result] Accrombessi M, Cook J, Dangbenon E, Yovogan B, Akpovi H, Sovi A, Adoha C, Assongba L, Sidick A, Akinro B, Osse R, Tokponnon F, Aikpon R, Ogouyemi-Hounto A, Padonou GG, Kleinschmidt I, Messenger LA, Rowland M, Ngufor C, Protopopoff N, Akogbeto MC. Efficacy of pyriproxyfen-pyrethroid long-lasting insecticidal nets (LLINs) and chlorfenapyr-pyrethroid LLINs compared with pyrethroid-only LLINs for malaria control in Benin: a cluster-randomised, superiority trial. Lancet. 2023 Feb 11;401(10375):435-446. doi: 10.1016/S0140-6736(22)02319-4. Epub 2023 Jan 24. PMID 36706778
- [Result] Sovi A, Yovogan B, Adoha CJ, Akinro B, Accrombessi M, Dangbenon E, Assongba L, Salako AS, Padonou GG, Messenger LA, Ngufor C, Cook J, Protopopoff N, Akogbeto MC. Efficacy of pyrethroid-pyriproxyfen and pyrethroid-chlorfenapyr nets on entomological indicators of malaria transmission: third year of a randomised controlled trial in Benin. Sci Rep. 2024 Jun 5;14(1):12958. doi: 10.1038/s41598-024-63883-2. PMID 38839981
- [Result] Ngufor C, Fagbohoun J, Fongnikin A, Ahoga J, Syme T, Ahogni I, Accrombessi M, Protopopoff N, Cook J, Dangbenon E, Sovi A, Baes M, Pigeon O, Todjinou D, Govoetchan R, Padonou GG, Akogbeto M. The attrition, physical and insecticidal durability of two dual active ingredient nets (Interceptor(R) G2 and Royal Guard(R)) in Benin, West Africa: results from a durability study embedded in a cluster randomised controlled trial. Parasit Vectors. 2024 Oct 7;17(1):420. doi: 10.1186/s13071-024-06504-1. PMID 39375740
- [Result] Accrombessi M, Cook J, Dangbenon E, Sovi A, Yovogan B, Assongba L, Adoha CJ, Akinro B, Affoukou C, Padonou GG, Kleinschmidt I, Messenger LA, Rowland M, Ngufor C, Akogbeto MC, Protopopoff N. Effectiveness of pyriproxyfen-pyrethroid and chlorfenapyr-pyrethroid long-lasting insecticidal nets (LLINs) compared with pyrethroid-only LLINs for malaria control in the third year post-distribution: a secondary analysis of a cluster-randomised controlled trial in Benin. Lancet Infect Dis. 2024 Jun;24(6):619-628. doi: 10.1016/S1473-3099(24)00002-1. Epub 2024 Feb 21. PMID 38401551
- [Derived] Sovi A, Adoha CJ, Yovogan B, Cross CL, Dee DP, Konkon AK, Sidick A, Accrombessi M, Ahouandjinou MJ, Osse R, Dangbenon E, Towakinou L, Agbangla C, Padonou GG, Churcher TS, Ngufor C, Cook J, Protopopoff N, Akogbeto MC, Messenger LA. The effect of next-generation, dual-active-ingredient, long-lasting insecticidal net deployment on insecticide resistance in malaria vectors in Benin: results of a 3-year, three-arm, cluster-randomised, controlled trial. Lancet Planet Health. 2024 Nov;8(11):e894-e905. doi: 10.1016/S2542-5196(24)00232-8. PMID 39515347